CLINICAL TRIAL: NCT04541290
Title: Tacrolimus as Treatment of Breast Cancer-Related Lymphedema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Gustaf Jørgensen, Doctor of Medicine, Principal investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tacrolimus_2020
Record Dates: First submitted 2020-08-28; First posted 2020-09-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Women with stage 1-2 lymphedema due to breast cancer treatment
  Interventions: Drug: Protopic 0.1 % Topical Ointment

INTERVENTIONS:
Drug: Protopic 0.1 % Topical Ointment — Applied in a thin layer covering all of the arm including the armpit and hand once a day for six months

SUMMARY:
BACKGROUND Breast cancer-related lymphedema is a severe and life-long side-effect to breast cancer treatment. The condition increases the risk of infections and decreases health-related quality of life (HR-QOL) in patients. No prophylactic or curative treatment is currently available for this condition.

CD4+-cells plays a critical role in the development of lymphedema. The cells facilitate inflammation and fibrosis formation in the subcutaneous tissue which inhibits lymphatic regeneration. Tacrolimus is an immunosuppressive and anti-inflammatory macrolide that targets the CD4+-cells. Tacrolimus as treatment of lymphedema has already shown promising results in animal studies. Tacrolimus has the potential to cure an otherwise uncurable and life-long side-effect of BC and will therefore benefit a large number of patients who suffers from BCRL.

AIM To assess the effect of Tacrolimus treatment on breast cancer-related lymphedema METHOD Study design A pilot study with a planned inclusion of 20 patients with a 12 month follow-up period. The purpose of this study is to assess the effect of tacrolimus treatment on lymphedema and HR-QOL. Results are attained from objective measures and questionnaires.

The patients will be seen at a consultation prior to the treatment start and then 3 times hereafter (at 3, 6 and 12 months) as follow up consultations where effect of treatment is evaluated.

Primary endpoint:

- Arm volume measured with water displacement test.

Secondary endpoints:

* Arm volume measured with measuring tape and calculated with volume of a cone formula
* Patient-reported outcome measured through the Danish versions of , LYMPH-ICF, DASH and SF-36 questionnaires
* Bioimpedance
* Lymphangiography Primary- and secondary endpoint data will be collected at each of the 3 consultations (prior to treatment and 3 and 6 months after the treatment start).

CLINICAL IMPACT This will be the first clinical pharmacological study on regarding treatment of lymphedema with Tacrolimus. This study will test the feasibility and efficacy of Tacrolimus ointment in a population of breast cancer patients who have developed lymphedema. The study may lead to a routine clinical implementation of tacrolimus ointment to patients diagnosed with Lymphedema. Regardless of the outcome, the study will benefit the patients and future research in the field of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-65 years
* Female
* Lymphedema diagnosis as a result of breast cancer treatment
* Active Lymphedema (excessive fluid)
* Significant lymphedema
* Grade I-II lymphedema
* Postmenopausal (Absence/lack of menstruation in at least 12 consecutive months) or continuously usage of contraceptive drugs (Spiral, birth-control pills, implant, transdermal patches, vaginal ring or depot injection). Contraceptive drugs must be used throughout the project and at least three weeks subsequent to the ending of the project (last application of the ointment).
* Clinically good general condition No lymphedema in the opposite arm (normal arm)
* Understands the purpose og the study and gives written consent to participate
* Can read and understand the danish language

Exclusion Criteria:

* Pregnant, breast-feeding or with wish of pregnancy within the next year
* Bilateral breast cancer
* Grade 0, III or IV lymphedema
* Known allergies for Tacrolimus or and other macrolide
* Removal of lymph nodes in the opposite armpit
* Suffers from psychiatric disorders that may affect the participation in the project
* Reduced kidney or liver function
* Defect skin-barrier
* Diagnosed immunodeficiency

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Change in Arm volume from Baseline | Baseline + change in arm volume at 3, 6 and 12 months from baseline
  measured with water displacement test. The patient lowers her arm in a basin of water (Bravometer, Novuqare BV, PJ Horst, NL) and arm volume is hereafter read in mL prior to and after the lowering of the arm. This method is established at the department we use for this project. Arm volume of both arms are measured at each consultation.

SECONDARY OUTCOMES:
Bioimpedance | Baseline + at 3, 6 and 12 month follow-up
  Bioimpedance measuring is a tool in estimating the excess liquid in the body. The test is non-invasive and is done by placing electrodes on the skin of the hands and feet similarly to the procedure of an ECG. Signals run through the electrodes connected to a machine that sends electric impulses trough the body and estimates the excess liquid in the extremities.
  The test is done at every consultation and has a duration of a couple of minutes. There is no side-effects or discomfort associated to the test.
Lymphangiography | Baseline + at 6 and 12 month follow-up
  An imaging-tool to quantify the lymph-flow and -vessels. ICG is a fluorescent that is absorbed in the lymphatic system and metabolized in the liver with a half-life at 3-4 minutes. The florescent ICG is detectable by cameras at specific wavelengths and is thereby possible to visualize. The outcome of this test is classified into groups: linear pattern and dermal backflow patterns. Dermal backflow patterns can then be subdivided into "splash", "stardust" and "diffuse patterns" via pattern-recognition.
  The procedure is done by injecting 0.02 mL ICG subcutaneously in the web space between each finger. Fluorescent imaging of the lymph-vessels and -flow is then obtained by using an infrared camera. There is no exposition of radiation associated with this test.
  The ICG lymphangiography is done on both arms. Outcome is measured as the pattern of the lymph-flow.
Questionnaire: Lymphedema Functioning, Disability and Health questionnaire (Lymph-ICF) LYMPH-ICF | Baseline + at 3, 6 and 12 month follow-up
  A Danish validated questionnaire developed specifically for lymphedema-patients. The questionnaire contains 5 domains: lymphedema symptoms, mental function, household activities, mobility activities movement and life and social activities.
  29 questions regarding the 5 domains are answered on a scale ranging from 0-10. Raw scores will be transformed into scores ranging from 0 (Worst) to 100 (best) using the original scoring key
Questionnaire: The disabilities of the arm, shoulder and hand (DASH) questionnaire | Baseline + at 3, 6 and 12 month follow-up
  A Danish validated questionnaire developed for patients with disabilities of the arms, shoulders and hands. It includes 38 questions about the patient's ability to perform different actions/movements. The questions are answered on a 5-step scale from not difficult to impossible.
  Raw scores will be transformed into scores ranging from 0 (Worst) to 100 (best) using the original scoring key
Questionnaire: 36-Item Short-Form Health Survey questionnaire (SF-36) | Baseline + at 3, 6 and 12 month follow-up
  A Danish validated generic quality of life-questionnaire. The questionnaire includes 36 questions regarding the patient's the general quality of life. The questions are answered on a 3-, 5- and 6-step scale and binary (Yes/No) depending on the question.
  Raw scores will be transformed into scores ranging from 0 (Worst) to 100 (best) using the original scoring key
Arm volume measured with measuring tape | Baseline + at 3, 6 and 12 month follow-up
  Manual measuring with measuring tape and then calculated with through volume of a cone formula

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD Prof. PhD, Study Chair — Department of Plastic Surgery at Odense University Hospital
Locations (1):
- Department of Plastic Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zou L, Liu FH, Shen PP, Hu Y, Liu XQ, Xu YY, Pen QL, Wang B, Zhu YQ, Tian Y. The incidence and risk factors of related lymphedema for breast cancer survivors post-operation: a 2-year follow-up prospective cohort study. Breast Cancer. 2018 May;25(3):309-314. doi: 10.1007/s12282-018-0830-3. Epub 2018 Feb 3. PMID 29397555
- [Background] Ribeiro Pereira ACP, Koifman RJ, Bergmann A. Incidence and risk factors of lymphedema after breast cancer treatment: 10 years of follow-up. Breast. 2017 Dec;36:67-73. doi: 10.1016/j.breast.2017.09.006. Epub 2017 Oct 6. PMID 28992556
- [Background] Grada AA, Phillips TJ. Lymphedema: Pathophysiology and clinical manifestations. J Am Acad Dermatol. 2017 Dec;77(6):1009-1020. doi: 10.1016/j.jaad.2017.03.022. PMID 29132848
- [Background] Taghian NR, Miller CL, Jammallo LS, O'Toole J, Skolny MN. Lymphedema following breast cancer treatment and impact on quality of life: a review. Crit Rev Oncol Hematol. 2014 Dec;92(3):227-34. doi: 10.1016/j.critrevonc.2014.06.004. Epub 2014 Jul 2. PMID 25085806
- [Background] Pusic AL, Cemal Y, Albornoz C, Klassen A, Cano S, Sulimanoff I, Hernandez M, Massey M, Cordeiro P, Morrow M, Mehrara B. Quality of life among breast cancer patients with lymphedema: a systematic review of patient-reported outcome instruments and outcomes. J Cancer Surviv. 2013 Mar;7(1):83-92. doi: 10.1007/s11764-012-0247-5. Epub 2012 Dec 5. PMID 23212603
- [Background] Terada M, Yoshimura A, Sawaki M, Hattori M, Naomi G, Kotani H, Adachi Y, Iwase M, Kataoka A, Sugino K, Mori M, Horisawa N, Ozaki Y, Iwata H. Patient-reported outcomes and objective assessments with arm measurement and bioimpedance analysis for lymphedema among breast cancer survivors. Breast Cancer Res Treat. 2020 Jan;179(1):91-100. doi: 10.1007/s10549-019-05443-1. Epub 2019 Sep 18. PMID 31535321
- [Background] Sackey H, Johansson H, Sandelin K, Liljegren G, MacLean G, Frisell J, Brandberg Y. Self-perceived, but not objective lymphoedema is associated with decreased long-term health-related quality of life after breast cancer surgery. Eur J Surg Oncol. 2015 Apr;41(4):577-84. doi: 10.1016/j.ejso.2014.12.006. Epub 2015 Jan 13. PMID 25659877
- [Background] Ghanta S, Cuzzone DA, Torrisi JS, Albano NJ, Joseph WJ, Savetsky IL, Gardenier JC, Chang D, Zampell JC, Mehrara BJ. Regulation of inflammation and fibrosis by macrophages in lymphedema. Am J Physiol Heart Circ Physiol. 2015 May 1;308(9):H1065-77. doi: 10.1152/ajpheart.00598.2014. Epub 2015 Feb 27. PMID 25724493
- [Background] Ogata F, Fujiu K, Matsumoto S, Nakayama Y, Shibata M, Oike Y, Koshima I, Watabe T, Nagai R, Manabe I. Excess Lymphangiogenesis Cooperatively Induced by Macrophages and CD4(+) T Cells Drives the Pathogenesis of Lymphedema. J Invest Dermatol. 2016 Mar;136(3):706-714. doi: 10.1016/j.jid.2015.12.001. Epub 2015 Dec 10. PMID 27015456
- [Background] Muller GG, Jose NK, de Castro RS, de Holanda EC. Long-term use of topical tacrolimus ointment: a safe and effective option for the treatment of vernal keratoconjunctivitis. Arq Bras Oftalmol. 2019 Mar-Apr;82(2):119-123. doi: 10.5935/0004-2749.20190026. Epub 2019 Jan 24. PMID 30698232
- [Background] Remitz A, Harper J, Rustin M, Goldschmidt WF, Palatsi R, van der Valk PG, Sharpe G, Smith CH, Dobozy A, Turjanmaa K; European Tacrolimus Ointment Study Group. Long-term safety and efficacy of tacrolimus ointment for the treatment of atopic dermatitis in children. Acta Derm Venereol. 2007;87(1):54-61. doi: 10.2340/00015555-0167. PMID 17225017
- [Background] Gardenier JC, Kataru RP, Hespe GE, Savetsky IL, Torrisi JS, Nores GD, Jowhar DK, Nitti MD, Schofield RC, Carlow DC, Mehrara BJ. Topical tacrolimus for the treatment of secondary lymphedema. Nat Commun. 2017 Feb 10;8:14345. doi: 10.1038/ncomms14345. PMID 28186091
- [Background] Harvey LA. REDCap: web-based software for all types of data storage and collection. Spinal Cord. 2018 Jul;56(7):625. doi: 10.1038/s41393-018-0169-9. No abstract available. PMID 29977003
- [Background] Lasinski BB, McKillip Thrift K, Squire D, Austin MK, Smith KM, Wanchai A, Green JM, Stewart BR, Cormier JN, Armer JM. A systematic review of the evidence for complete decongestive therapy in the treatment of lymphedema from 2004 to 2011. PM R. 2012 Aug;4(8):580-601. doi: 10.1016/j.pmrj.2012.05.003. PMID 22920313
- [Background] Damstra RJ, Glazenburg EJ, Hop WC. Validation of the inverse water volumetry method: A new gold standard for arm volume measurements. Breast Cancer Res Treat. 2006 Oct;99(3):267-73. doi: 10.1007/s10549-006-9213-0. Epub 2006 Jun 3. PMID 16752072
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Klassen AF, Dominici L, Fuzesi S, Cano SJ, Atisha D, Locklear T, Gregorowitsch ML, Tsangaris E, Morrow M, King T, Pusic AL. Development and Validation of the BREAST-Q Breast-Conserving Therapy Module. Ann Surg Oncol. 2020 Jul;27(7):2238-2247. doi: 10.1245/s10434-019-08195-w. Epub 2020 Jan 21. PMID 31965369
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123
- [Derived] Gulmark Hansen FC, Jorgensen MG, Sorensen JA. Treatment of Breast Cancer-Related Lymphedema With Topical Tacrolimus: A Prospective, Open-Label, Single-Arm, Phase II Pilot Trial. J Breast Cancer. 2023 Feb;26(1):46-59. doi: 10.4048/jbc.2023.26.e2. Epub 2023 Jan 19. PMID 36762782
- See also: NORDICAN. Association of the Nordic Cancer Registries. Danish Cancer Society. Available from http://www.ancr.nu, accessed on 24 February 2020. Cancer [Internet]. 2011;1-2. — http://www-dep.iarc.fr/NORDCAN/english/frame.asp
- See also: Tacrolimus Topical: MedlinePlus Drug Information [Internet]. [cited 2020 Feb 24]. — http://www.medlineplus.gov/druginfo/meds/a602020.html